CLINICAL TRIAL: NCT06987383
Title: Vibegron - A Novel Treatment for Multisystem Functional Decline in Aging and Obesity
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Brinkley.Vibegron; R21AG091075 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Vibegron; aging; metabolism; physical function; cognitive function
MeSH Terms: conditions — Obesity | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pharmacy will provide Vibegron tablets and create matching placebo. Participants will be randomized 1:1 to either arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibegron (Experimental): Participants in this arm will take 75mg/day Vibegron for 12 weeks.
  Interventions: Drug: Vibegron
- Placebo (Placebo Comparator): Participants in this arm will take placebo daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vibegron — A drug in a class of medications called beta-3 adrenergic agonists; approved for use with Overactive Bladder; 75mg tablets will be used in this study
  Other Names: Gemtesa
  Arms: Vibegron
Drug: Placebo — Tablets made of inert substance that looks like the vibegron tablets but has no therapeutic value
  Arms: Placebo

SUMMARY:
This 12-week randomized, double-blind, placebo-controlled trial will test the hypothesis that Vibegron (brand name GEMTESA) can improve energy metabolism, cardiometabolic risk factors, and physical and cognitive function in middle-aged and older adults with obesity.

DETAILED DESCRIPTION:
Aging is characterized by the gradual loss of physiological integrity, and this process may be accelerated in the presence of obesity, increasing susceptibility to disease, frailty, and death. Although the shared molecular pathways involved have not been fully elucidated, adipose tissue dysfunction is likely a key contributor to multisystem functional decline in aging and obesity. Despite growing evidence that β3 adrenergic receptor (β3AR) mediated activation of brown adipose tissue (BAT) may alter pathophysiological pathways implicated in various aging-related diseases including metabolic, cardiovascular, and neurodegenerative diseases, BAT has been largely ignored in aging research. This study will randomize 40 middle-aged and older adults (45-75 yrs) with obesity to the β3AR agonist Vibegron (75 mg/day) or placebo for 12 weeks to compare their effects on various bioenergetic, cardiometabolic, physical function, and cognitive outcomes. Potential study candidates will be screened by telephone to determine basic interest and eligibility. Individuals who pass this initial screening will then undergo an in-person screening at Atrium Health Wake Forest Baptist. Enrolled participants will be randomized 1:1 to Vibegron or placebo and will be instructed to take the study drug by mouth once daily for 12 weeks. Study outcomes will be assessed at the baseline and follow-up visits and at one safety/compliance visit. Participants will self-report demographic, behavioral, and medical information using questionnaires. They will also complete functional tests to assess muscle strength/power and mobility, DXA and CT scans to assess body composition and body fat distribution, and remote monitoring to assess core body temperature. In addition, participants will have their blood drawn for the assessment of glucose/insulin and lipid indices, for screening and safety purposes, and for storage of plasma/serum samples. Blood samples will also be used to assess mitochondrial bioenergetics in peripheral blood mononuclear cells and thermogenic and adipokine protein expression in adipose tissue-derived small extracellular vesicles. Safety will be assessed based on treatment-related adverse events and measurement of blood chemistries and vitals. To assess medication adherence, participants will be instructed to keep a daily dosing diary and to bring the log, along with empty pill bottles, to the safety/compliance visit for review by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI ≥30 kg/m2 or BMI ≥27 kg/m2 with a waist circumference >102 cm for men and >88 cm for women)

Exclusion Criteria:

* Body weight ≥450 pounds
* Major depression
* Evidence of cognitive impairment
* Uncontrolled diabetes (hemoglobin A1c >7%)
* Weight gain or loss of ≥5% over the past 6 months
* Prior weight loss procedure (e.g., gastric bypass, sleeve gastrectomy, gastric banding)
* Regular use of the following: weight loss medications (e.g., Orlistat, Belviq, Contrave, Saxenda, Phentermine, Qsymia); medications or dietary supplements known to alter energy metabolism; adrenergic agonists or beta blockers
* Symptoms of urinary retention, incontinence, urgency, and frequency or current use of an antimuscarinic medication to treat overactive bladder
* Benign prostate hyperplasia
* Significant medical illness or organ failure, such as uncontrolled hypertension, advanced kidney disease, liver disease, thyroid disease, or active neoplastic disease
* Diagnosis of a neurodegenerative illness (e.g., mild cognitive impairment, dementia, Parkinson's disease, Multiple Sclerosis)
* History of a clinically significant stroke
* Cardiac arrhythmia or an abnormal Electrocardiogram
* Drug/substance abuse or excessive alcohol use within the past 6 months
* Contraindication to Vibegron or any of its components
* Current participation in another intervention or research study that prohibits co-enrollment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Resting Metabolic Rate | Baseline
  Resting metabolic rate (RMR) will be measured by indirect calorimetry using a computerized metabolic cart that provides valid and reliable measurement of oxygen consumption and carbon dioxide production - RMR can be estimated using formulas such as the Mifflin-St Jeor equation:
  Males: RMR = 10 * weight (kg) + 6.25 * height (cm) - 5 * age (years) + 5 Females: RMR = 10 * weight (kg) + 6.25 * height (cm) - 5 * age (years) - 161
Resting Metabolic Rate | Week 12
  Resting metabolic rate (RMR) will be measured by indirect calorimetry using a computerized metabolic cart that provides valid and reliable measurement of oxygen consumption and carbon dioxide production - RMR can be estimated using formulas such as the Mifflin-St Jeor equation:
  Males: RMR = 10 * weight (kg) + 6.25 * height (cm) - 5 * age (years) + 5 Females: RMR = 10 * weight (kg) + 6.25 * height (cm) - 5 * age (years) - 161

SECONDARY OUTCOMES:
Glucose Tolerance Level | Baseline and Week 12
  Glucose tolerance will be assessed using a standard 75-g oral glucose load to measure changes in glucose and insulin levels. Glucose tolerance will be defined as the 2-hour glucose level - a normal two-hour post-glucose level is below 140 mg/dL (7.8 mmol/L). Levels between 140 and 199 mg/dL (7.8 and 11 mmol/L) indicate impaired glucose tolerance (also called prediabetes), while levels of 200 mg/dL (11.1 mmol/L) or higher suggest diabetes.
Expanded Short Physical Performance Battery (eSPPB) | Baseline and Week 12
  Lower extremity function will be assessed using the eSPPB which measures balance, gait speed, and leg strength - Each component is scored separately, and then the scores are summed to give a total score ranging from 0 (worst) to 12 (best) - The total score is calculated by summing the scores from the three subtests.
  A higher total score indicates better lower extremity function, while a lower score indicates more functional limitations.

OTHER OUTCOMES:
Core body temperature | Baseline and Week 12
  Core body temperature will be measured continuously using a temperature monitoring patch worn on the chest.
Lipid levels | Baseline, Week 4, and Week 12
  Plasma levels of total cholesterol, VLDL cholesterol, HDL cholesterol, and triglycerides will be measured in fasted blood samples.
Depressive Symptoms: 15-item Geriatric Depression Scale (GDS-15) | Baseline and Week 12
  Questionnaire used to measure depressive symptoms in the elderly; ranges from 0-15 with higher scores indicating greater severity of depression; score of 0-4 is within normal range; score of 5-8 mild depression; score of 9-11 moderate depression; score of 12-15 severe depression
Quality of Life: Medical Outcomes Study Short Form 36 (SF-36) | Baseline and Week 12
  Quality of life questionnaire with a score that ranges from 0 to 100 with higher scores indicating better quality of life.
Compliance Rate | Baseline, Week 4, and Week 12
  Compliance will be defined based on the number of daily doses taken relative to the total number of doses prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Tina E Brinkley, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No